CLINICAL TRIAL: NCT01290588
Title: Aqueous Humor Dynamics and Biometric Parameters in Eyes of Children
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0364-09-FB
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children of Caucasian descent: Healthy children of Caucasian descent.
- Adults of Caucasian descent: Healthy adult eyes of Caucasian descent.
- Children of African-American descent: Healthy children of African-American descent.
- Adults of African-American descent: Healthy adults of African-American descent.

SUMMARY:
The purpose of this study is to determine the effect of age and ethnic background on ocular aqueous humor dynamics and biometric parameters. Data of normal healthy children and adults will be used as controls for future study of juvenile glaucoma, and diabetes and potentially for any other condition that affects intraocular pressure in children.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy and a leading cause of blindness in the United States1 and the second leading cause of blindness worldwide. In glaucoma, vision is lost through apoptosis of retinal ganglion cells. Diagnosis of glaucoma is usually based on a combination of progressive, characteristic vision loss (measured using visual field testing) and progressive optic nerve head damage (as detected through dilated fundus examinations or optic disc photography). While ocular hypertension (OHT) is not sufficient for a diagnosis of glaucoma, it is the greatest prognostic and modifiable factor. In fact, the only effective treatment for glaucoma currently is to treat the elevated IOP. This treatment does not provide a cure but it does slow glaucoma progression. IOP is determined by the balance between aqueous production (flow) and aqueous humor outflow through either the trabecular meshwork or uveoscleral pathway. Therefore, all clinically available glaucoma treatments are designed to increase drainage and/or reduce production. The main purpose of the current study is the determination of aqueous humor dynamics.

There are two main types of glaucoma, "open angle" or chronic glaucoma and "closed angle" or acute glaucoma. Open angle glaucoma tends to progress slowly and may remain undetected until the patient notices a change in vision. On the other hand, angle closure glaucoma appears suddenly and can be very painful, therefore is often diagnosed more quickly. The chance of suffering from either one of these types of glaucoma depends greatly on one's ethnic background. People suffering from primary angle-closure glaucoma (PACG) have short axial lengths and shallow anterior chambers. These physical dimensions are found predominantly in people from Asia and India. Angle-closure glaucoma is caused by factors that either pull or push the iris up into the angle, physically blocking the drainage of aqueous humor and increasing the resistance to outflow. The IOP will increase to dangerous levels in order to drain the fluid through the obstructed outflow pathways.

Narrow angles are not present in children. As a person ages, the lens of the eye continues to grow. In some but not all people, this growth pushes the iris forward, narrowing the angle. Risk factors for developing narrow angles include Asian ethnicity, hyperopia, family history, and advanced age. Prevalence figures identify East Asia as home to the majority of those affected by PACG. PACG is acknowledged as a major cause of ocular morbidity in Chinese populations and is more common among Chinese people than among Caucasian people. Part of the global project is to travel to China to study Chinese children and adults. This will be done in collaboration with Ganzu Hospital in Lanzhou, China. This is not part of the current protocol.

Open angle glaucoma typically occurs in older patients in the sixth decade of life or more. African-Americans have up to six times higher risk of developing the condition than the general population especially if there is a family history of glaucoma. Additionally, patients who are highly myopic, have diabetes mellitus, or have cardiovascular problems are at high risk of developing open angle glaucoma. Visual acuity, axial length and medical history will be collected as part of the current protocol.

Unlike narrow angle glaucoma, patients with open angle glaucoma have a gradual blockage of aqueous humor outflow despite a seemingly open chamber angle in the drainage pathway. As the eye ages, the drainage system can become clogged with debris causing pressure inside the eye to build to harmful levels. Open angle glaucoma can develop gradually and remain undetected for years. Because there is usually no pain experienced over the months or years of development and no other symptoms are apparent, the patient is often unaware of the existence of this serious eye disorder. Since African-Americans are at such a high risk for contracting glaucoma, children and adults of this ethnic background will be included in this study.

Glaucoma can occur in children as well as adults. Glaucoma that begins before the child is 3 years old is called infantile or congenital glaucoma. Glaucoma manifesting itself in a child's teens is juvenile glaucoma. There are many causes of childhood glaucoma, such as heredity, or injury or certain eye disorders. Once the investigators collect information on aqueous humor dynamics in healthy teenaged children, the investigators will study children of the same age with glaucoma. The investigators are planning to conduct these studies at Paracelsus University in Salzburg Austria. That is not part of the present protocol.

In the recent rabbit study, the investigators have learned that there are distinctive circadian rhythms of IOP and aqueous humor dynamics in juvenile and adult rabbits. In the ongoing clinical study of ocular hypertensive patients, the investigators are finding that some glaucoma medications are not effective at night despite being efficacious during the day. This has significant clinical importance. The investigators are including the study of aqueous humor dynamics at night in the current protocol to determine the normal circadian patterns for each ethnic group and age group.

In animal studies, the investigators have found that there are several significant differences in aqueous humor dynamics in immature animals compared to adult animals. This is not just a continuum of changes occurring between young and old adults. The investigators predict that important changes also take place in the ocular fluid dynamics of the eye as a child matures. The major changes may occur during puberty. Understanding normal ocular physiology in children will help us to understand the pathological changes taking place in juvenile glaucoma. The clinical importance of this project is immense

ELIGIBILITY:
Inclusion Criteria:

* Subjects must not have any ocular diseases
* Children, 15 - 18 years of age
* Adults, 30 - 50 years of age

Exclusion Criteria:

* Women who are pregnant or lactating
* Aphakia or pseudophakia
* Chronic or recurrent severe ocular inflammatory disease.
* Ocular infection or inflammation within three (3) months of screening visit.
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Any abnormality preventing reliable tonometry of either eye.
* History of any ocular pathology (including dry eye).
* A cup-to-disc ratio greater than 0.8
* History of intraocular surgery
* History of ocular laser surgery
* History of hypersensitivity or allergy to beta blockers and sulfa drugs.
* History of severe, unstable or uncontrolled cardiovascular, hepatic or renal disease.
* History of bronchial asthma or chronic obstructive pulmonary disease (COPD).
* Inability to discontinue contact lens wear.
* Diagnosis of ocular hypertension or glaucoma or any ocular disease

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Children
  * Adults
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol B Toris, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmology and Visual Sciences, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No